CLINICAL TRIAL: NCT02933216
Title: Comparison of the Therapeutic Effects of Vaginal Repair and Hysteroscopic Combined With Laparoscopic Excision in the Treatment of Cesarean Scar Diverticula
Brief Title: Comparison of the Therapeutic Effects of VR and Hysteroscope + Laparoscope in the Treatment of Cesarean Scar Diverticula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSD-002
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cesarean Scar Diverticula
Keywords: Cesarean Scar Diverticula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- VR: The CSD patients are received treatment of vaginal repair.
- hysteroscope + laparoscope: The CSD patients are received treatment of hysteroscopic combined with laparoscopic excision.

SUMMARY:
Cesarean scar diverticula (CSD) is a novel recognized cause of postmenstrual abnormal uterine bleeding in women. No clinical guidelines have been issued for the management of CSD. Currently, several limited surgical management procedures for CSD have been reported, such as hysteroscopic combined with laparoscopic excision (abbreviated as hysteroscope + laparoscope) and vaginal repair of CSD (abbreviated as VR). However, which management can achieve better clinical effects remains unknown. Therefore, this prospective study is designed to compare the therapeutic effects between VR and hysteroscope + laparoscope in the treatment of CSD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are younger than 40.
2. Clearly diagnosed with CSD.
3. Experiencing clinical features of abnormal uterine bleeding, prolonged menstrual flow (the duration of menstruation is more than 7 days).
4. The thickness of the remaining muscular layer of CSD was less than 3 mm.
5. The women are at least 20 years old with singleton pregnancies and had undergone a cesarean delivery after at least 37 weeks of gestation.
6. The medicine conservative treatment is invalid.
7. Refusing or use birth control pills contraindications.
8. No serious medical problems (important viscera function in the normal range).
9. No uterine fibroids, endometriosis, adenomyosis, and patients with ovarian cysts.
10. No gynaecology or other malignant tumors.
11. Sign the informed consent.

Exclusion Criteria:

1. Over the age of 40;
2. Indefinite diagnosis.
3. The absence of clinical manifestations of CSD.
4. The presence of menstrual irregularities before cesarean delivery.
5. Coagulation disorders.
6. Malignant tumors.
7. With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
8. Known chronic inflammatory diseases, any other uterine diseases (such as uterine fibroids, endometriosis and adenomyosis), uterine surgery except cesarean section.
9. Use of intrauterine devices.
10. Unwilling to comply with the research plan.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cesarean section diverticula patients from Nov 2016 until June 2018 in Shanghai First Maternity and Infant Hospital, Tongji University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
thickness of the remaining muscular layer (mm) | 6 months after surgery
  The thickness of the remaining muscular layer is measured by transvaginal ultrasound.

SECONDARY OUTCOMES:
duration of menstruation (day) | 6 months after surgery
  The menstruation duration in CSD patients is collected 6 months after surgery.
the length of CSD (mm) | 6 months after surgery
  The length of CSD is measured by transvaginal ultrasound.
the depth of CSD (mm) | 6 months after surgery
  The depth of CSD is measured by transvaginal ultrasound.
the width of CSD (mm) | 6 months after surgery
  The width of CSD is measured by transvaginal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, M.D., Ph.D.,, Study Chair — Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University
Locations (1):
- Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China